CLINICAL TRIAL: NCT03275779
Title: Investigating the Role of Resistance Exercise Frequency in the Regulation of Skeletal Muscle Mass
Acronym: EXFREQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ERN_17-0997
Record Dates: First submitted 2017-08-31; First posted 2017-09-08 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-12

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Frequency Condition (Experimental): Participants complete 7 days of habitual physical activity followed by a 7 day period where participants complete a single bout of unilateral resistance exercise.
  Interventions: Behavioral: Low Frequency Condition
- High Frequency Condition (Experimental): Participants complete 7 days of habitual physical activity followed by a 7 day period where participants complete the same total volume of resistance exercise as the low frequency condition as five smaller bouts of unilateral resistance exercise.
  Interventions: Behavioral: High Frequency Condition

INTERVENTIONS:
Behavioral: Low Frequency Condition — Young, untrained participants complete 7 days of habitual physical activity followed by a 7 day period where participants complete a single bout of unilateral resistance exercise.
  Arms: Low Frequency Condition
Behavioral: High Frequency Condition — Young, untrained participants complete 7 days of habitual physical activity followed by a 7 day period where participants complete the same total volume of resistance exercise as the low frequency condition as five smaller bouts of unilateral resistance exercise.
  Arms: High Frequency Condition

SUMMARY:
This study will investigate whether manipulating resistance exercise frequency impacts muscle protein synthesis rates. The investigators will test the hypothesise that a higher resistance exercise frequency will result in greater muscle protein synthesis rates than a lower resistance exercise frequency.

DETAILED DESCRIPTION:
Resistance exercise is currently the most effective means of building or maintaining muscle mass. Resistance exercise guidelines generally suggest that those looking to increase muscle mass should train each muscle group once to twice per week. However, it has been proposed that it may be of greater benefit to train a muscle group with a higher frequency (i.e., four to six times per week) than currently suggested. If true, completing the same total volume of resistance exercise in more frequent, smaller bouts could prove to be a more beneficial strategy to optimally build or maintain muscle mass.

Therefore, this study will investigate whether manipulating resistance exercise frequency impacts cumulative muscle protein synthesis rates in young individuals. Participants will undergo a 7 day period of habitual activity before completing the same total volume of resistance exercise as either; i) one isolated bout (low frequency) or ii) five smaller bouts (high frequency) over a period of 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (18.5-29.99 kg/m2)
* Untrained - defined as: Perform activities of daily living and recreation but have completed no regular lower body resistance-type exercise (e.g., weight training) activity in the last year.
* Good general health

Exclusion Criteria:

* Lidocaine allergy
* Hypertension (≥140/90 mmHg)
* Current participation in another clinical study
* Previous participation in this study
* Bleeding disorder/s
* Current or recent smoker
* Vegetarian or vegan
* Past history of substance abuse and/or taking prescription or non-prescription medication (e.g., beta-blockers, insulin or thyroxine) or supplements that may influence normal metabolic responses.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants must be male.
Enrollment: 9 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Change in muscle protein synthesis (FSR %/day) | At day 10 and 15.
  The change in muscle protein synthesis rates (FSR %/day) from baseline will be determined between the low and high frequency conditions at days 10 and 15 using deuterium oxide (D2O).

SECONDARY OUTCOMES:
Change in satellite cell response | At day 10 and 15.
  The change in acute satellite cell response will be determined in muscle samples following low and high frequency resistance exercise at days 10 and 15.

CONTACTS AND LOCATIONS:
Overall Officials: Gareth Wallis, PhD, Principal Investigator — University of Birmingham
Locations (1):
- School of Sport Exercise and Rehabilitation Sciences, University of Birmingham, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No